CLINICAL TRIAL: NCT05960656
Title: Protocol l: SGLT2 Inhibitors, Ketogenesis, and Ketoacidosis
Brief Title: SGLTi, Hepatic Glucose Production and Ketogenesis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSC20230457H - 440509; R01DK024092 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Pancreatic clamp; Endogenous glucose production; Ketogenesis; Gluconeogenesis; Lipolysis; Norepinephrine turnover
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A randomized controlled 2 arm clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomly assigned 2:1 active drug:placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 25 mg/day
  Interventions: Drug: Empagliflozin 25 MG
- Placebo/Control Group (Placebo Comparator): Placebo control
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — A medication used in the management and treatment of type 2 diabetes mellitus. It is in the sodium-glucose co-transporter (SGLT-2) class of medications.
  Other Names: Jardiance
  Arms: Empagliflozin
Other: Placebo — Inert tablet
  Other Names: Placebo for empagliflozin
  Arms: Placebo/Control Group

SUMMARY:
In this study, we will test the hypothesis that distinct mechanisms account for the SGLT2i-induced stimulation of ketogenesis and lipolysis versus endogenous (hepatic) glucose production in patients with type 2 diabetes (T2D) and type 1 diabetes (T1D), and that the increases in ketone production and lipolysis can be prevented by concomitant administration of the thiazolidinedione pioglitazone. We will conduct five distinct experiments to test this hypothesis in patients with T2D and T1D.

MAIN STUDY: To examine the effect of empagliflozin versus empagliflozin/pancreatic clamp on EGP (6,6, D2-glucose), gluconeogenesis (D2O), lipolysis (U-2H-glycerol), ketogenesis (13C-palmitate conversion to 3-betahydroxybuyrate), and norepinephrine turnover (3H-NE) in type 2 diabetes subjects.

DETAILED DESCRIPTION:
MAIN STUDY

Participants: 30 T2D subjects, age = 30-75 y, BMI = 23-38 kg/m2, HbA1c = 7.0-11%, eGFR > 60 ml/min/1.73m2, BP < 160/90 mmHg. Participants must be in general good health based on medical history, physical exam, screening blood chemistries, CBC, TSH/T4, EKG, and urinalysis. Patients must have stable body weight (±1.5 kg) over the last 3 months and must not participate in an excessively heavy exercise program. Patients treated with diet, SU, metformin, or SU/MET are eligible. Patients treated with GLP-1 RA, DPP-4i, TZD, or insulin are excluded. Patients taking medications (other than SU/MET) known to affect glucose metabolism are excluded. Statin therapy is permissible if the dose has been stable for at least 3 months. Subjects with evidence of proliferative retinopathy or eGFR < 60 are excluded. Women of childbearing potential are excluded unless they are taking/using appropriate contractive medications/devices.

Protocol: Subjects will be randomized to receive empagliflozin (n=20) or placebo (n=10) in 2:1 ratio. Subject stratification will be done according to the following parameters: age (> or < 50 y), BMI (> or < 30 kg/m2), eGFR (> or < 80 ml/min/1.73 m2), HbA1c (> or < 8.5%). Each subject will participate in two studies performed in random order with 7-10 day interval between studies. In Study 1a, EGP will be measured with a prime-continuous 6,6, D2-glucose infusion and lipolysis will be measured with prime-continuous infusion of U-2H-glycerol. The rate of ketogenesis will be determined by infusion of 13C palmitate and quantitating the enrichment of 13C in 3-hydroxybutyrate (BHB). Total body NE turnover will be measured with 3H-norepinephrine (3H-NE) infusion before and after empagliflozin administration. Study 1b will be similar to Study 1a with one exception. EGP, lipolysis, and ketogenesis, and NE turnover will be measured under pancreatic clamp conditions.

ELIGIBILITY:
Patients with T2D

Inclusion Criteria:

* Ages 30-75 years
* Body Mass Index (BMI) 21-45 kg/m2
* Hemoglobin A1C (HbA1c) = 7.0-11%
* Estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m2
* Blood Pressure (BP) < 160/90 mmHg
* Participants must be in general good health based on medical history, physical exam, screening blood chemistries, complete blood chemistry (CBC), thyroid stimulating hormone/thyroxine (TSH/T4), electrocardiogram (EKG), and urinalysis
* Stable body weight (±1.5 kg) over the last 3 months and must not participate in an excessively heavy exercise program
* Patients treated with diet, sulfonylurea (SU), metformin (MET), or SU/MET
* Statin therapy is permissible if the dose has been stable for at least 3 months

Exclusion Criteria:

* Patients treated with Glucagon-like peptide 1 receptor agonists (GLP-1 RA), Dipeptidyl Peptidase IV inhibitors (DPP-4i), Thiazolidinediones (TZD), or insulin are excluded
* Patients taking medications (other than SU/MET) known to affect glucose metabolism are excluded
* Subjects with evidence of proliferative retinopathy or eGFR < 60 are excluded
* Women of childbearing potential are excluded unless they are taking/using appropriate contractive medications/devices

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Endogenous Glucose Production (EGP) | 0 and 300 minutes
  Measurement of Endogenous Glucose Production (EGP) using stable isotope (6,6, D2- glucose infusion).

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute/UH, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with NIH and as a publication in a peer reviewed journal once data are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study end after analysis of data.